CLINICAL TRIAL: NCT07098949
Title: Multicenter Randomized Controlled Clinical Study on Acupuncture Combined With Adjuvant Chemotherapy for the Prevention of Recurrence and Metastasis After Gastric Cancer Surgery
Brief Title: Acupuncture Combined With Chemotherapy for Gastric Cancer After Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024ZD0521302; 2024ZD0521302 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-07-14; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Accupuncture; Adjuvant chemotherapy; Recurrence
MeSH Terms: conditions — Stomach Neoplasms; Recurrence | interventions — Acupuncture Therapy; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Treatment Group (Experimental): Acupuncture for three times every 3 weeks(once a week, one cycle of adjuvant chemotherapy), a total of 4 cycles of adjuvant chemotherapy.
  Interventions: Other: Acupuncture; Drug: Chemotherapy
- Sham Acupuncture Group (Sham Comparator): Sham acupuncture procedure at the same acupoints and treatment schedule as the acupuncture group, utilizing a blunt-tipped sham needle for superficial pressure.
  Interventions: Other: Sham Acupuncture; Drug: Chemotherapy

INTERVENTIONS:
Other: Acupuncture — The patient takes a sitting or lateral position. The following acupoints are selected Baihui (GV20), Yintang (EX-HN3), Zhongwan (CV12), Bilateral Neiguan (PC6), Bilateral Zusanli (ST36), Bilateral Sanyinjiao (SP6), Bilateral Gongsun (SP4), Bilateral Pishu (BL20). Electroacupuncture is applied at bilateral Sanyinjiao (SP6) and bilateral Zusanli (ST36) by connecting them to an electroacupuncture device. The needles are retained for 30 minutes.
  Arms: Acupuncture Treatment Group
Other: Sham Acupuncture — sham acupuncture procedure that mirrors the acupuncture treatment in terms of acupoint selection and treatment schedule. However, instead of actual needle insertion, a blunt-tipped sham needle will be used to apply superficial pressure at the designated acupoints. The design of the sham needle includes a base that allows for simulated insertion, providing patients with a mild sensation of pressure and a visual cue as the needle appears to move toward the skin. This innovative approach ensures that while participants experience a similar tactile sensation, there is no penetration of the skin, distinguishing it clearly from the actual acupuncture treatment.
  Arms: Sham Acupuncture Group
Drug: Chemotherapy — Adjuvant chemotherapy with either the XELOX (capecitabine + oxaliplatin) or SOX (S-1 + oxaliplatin) regimen

SUMMARY:
This multicenter, randomized, parallel-group clinical trial aims to evaluate the efficacy of acupuncture combined with adjuvant chemotherapy in patients with gastric cancer who have undergone surgery. Participants will be randomly assigned in a 1:1 ratio to receive either acupuncture or sham acupuncture during the adjuvant chemotherapy period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with gastric cancer who have undergone R0 resection of the stomach/ distal stomach with D2 lymphadenectomy and are planned to receive postoperative adjuvant chemotherapy
2. Postoperative pathological diagnosis of gastric cancer, with pathological staging of pII/pIII (American Joint Committee on Cancer, AJCC)
3. No recurrence or metastasis confirmed by imaging examination
4. Performance Status (PS) score of 0-2
5. Age between 18 and 75 years
6. Normal bone marrow, liver, and kidney function:

   * Normal bone marrow function: Neutrophil count ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90g/L
   * Normal kidney function: Serum creatinine ≤1.5mg/dl (133μmol/L) and/or creatinine clearance ≥60ml/min
   * Normal liver function: Total serum bilirubin level ≤1.5 times the upper limit of normal (ULN), serum aspartate aminotransferase (AST) & alanine aminotransferase (ALT) ≤2.5 times ULN
7. Signed informed consent, and the patient voluntarily accepts treatment according to this protocol

Exclusion Criteria:

1. Unable to complete baseline assessment
2. Individuals with a fear of acupuncture
3. Those planning to receive postoperative adjuvant radiotherapy
4. History of blood system diseases, organ transplant history, or those requiring long-term oral immunosuppressants
5. Individuals with implanted cardiac pacemakers
6. Those who have received acupuncture treatment within the past 6 weeks
7. Fever within 3 days prior to enrollment with a temperature above 38°C or clinically significant infections(Subject to enrollment once infection is managed)
8. Currently receiving or having used the investigational drug or device within 4 weeks prior to the first intervention of the study
9. Presence of other primary tumors
10. Pregnant or breastfeeding women, individuals with mental illness, intellectual or language disabilities, those lacking legal capacity, or those whose medical or ethical reasons affect the continuation of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From the date of surgery until the date of first documented tumor recurrence, distant metastasis, or death from any cause, whichever occurs first, assessed up to 5 years.

SECONDARY OUTCOMES:
Average trajectory of FACT-Gastric TOI over time | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. FACT-Gastric TOI is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS) of the FACT-Gastric Scoring. The range of FACT-Gastric TOI is 0-132. The higher the score, the better the quality of life.
Total AUC of FACT-Gastric TOI | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. FACT-Gastric TOI is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS) of the FACT-Gastric Scoring. The range of FACT-Gastric TOI is 0-132. The higher the score, the better the quality of life. The area under curve (AUCs) are calculated by linear interpolation respectively, and then added together for the total AUC during the 4 cycles of chemotherapy.
Average trajectory of GASTRIC CANCER SUBSCAL (GaCS) of FACT-Gastric | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  The GaCS of FACT-Gastric focuses on the symptoms and functions related to gastric cancer specifically. The range of GaCS is 0-76. The higher the score, the better the quality of life.
Total AUC of GASTRIC CANCER SUBSCAL (GaCS) of FACT-Gastric | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  The GaCS of FACT-Gastric focuses on the symptoms and functions related to gastric cancer specifically. The range of GaCS is 0-76. The higher the score, the better the quality of life. The area under curve (AUCs) are calculated by linear interpolation respectively, and then added together for the total AUC during the 4 cycles of chemotherapy.
Average trajectory of FACT-Gastric Scoring over time | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. It is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, SOCIAL WELL BEING (SWB) SUBSCALE, EMOTIONAL WELL BEING (EWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS). The range of FACT-Gastric scoring is 0-184. The higher the score, the better the quality of life.
Total AUC of FACT-Gastric Scoring | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. It is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, SOCIAL WELL BEING (SWB) SUBSCALE, EMOTIONAL WELL BEING (EWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS). The range of FACT-Gastric scoring is 0-184. The higher the score, the better the quality of life. The area under curve (AUCs) for each cycle are calculated by linear interpolation respectively, and then added together for the total AUC during the 4 cycles of chemotherapy.
Average trajectory of Modified Edmonton Symptom Assessment Scale | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  Edmonton symptom assessment scale (ESAS) is a questionnaire used for symptom assessment in cancer patients. It was composed of 10 items with score range of 0-10 for each item, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, shortness of breath, and other. ESAS was then modified in 2015, with additional symptoms of constipation and sleep. The higher the score, the worse the symptom is.
Total AUC of Modified Edmonton Symptom Assessment Scale | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  Edmonton symptom assessment scale (ESAS) is a questionnaire used for symptom assessment in cancer patients. It was composed of 10 items with score range of 0-10 for each item, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, shortness of breath, and other. ESAS was then modified in 2015, with additional symptoms of constipation and sleep. The higher the score, the worse the symptom is.The AUCs are calculated by linear interpolation respectively, and then added together for the total AUC during the 4 cycles of chemotherapy.
Overall survival | From the date of surgery until the date of death from any cause, assessed up to 5 years.
Chemotherapy completion rate | The number of patients who have received 8 Cycle chemotherapy divided by the total number of patients in each group, assessed up to 8 months.
  Record the course and dosage of adjuvant chemotherapy for patients and calculate the chemotherapy completion rate.
Traditional Chinese Medicine Symptom Assessment | Assessed at baseline (Day1 at randomization), the first week of each Cycle 1-4 (each cycle is 21 days), the first day of Cycle 5 (each cycle is 21 days), and the time of recurrence or metastasis identified through CT/MRI imaging diagnosis
  The MDASI-TCM scale was evaluated before chemotherapy

OTHER OUTCOMES:
Traditional Chinese medicine syndrome data | Assessed on the last day of each chemotherapy cycle (each cycle is 21 days), up to treatment completion (maximum 8 cycles).
  The scale evaluates symptoms (e.g., fatigue, poor appetite) scored 0-10 per item. Scores are collected by TCM physicians and reported as mean change from baseline
Adverse events | Assessed within 1 day prior to each cycle of chemotherapy ( 21 days per cycle), up to treatment completion (maximum 8 cycles).
  Incidence of treatment-related adverse events (TRAEs) graded by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Prof, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (3):
- China (3):
  - The first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Sixth Affiliated Hospital ,Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol